CLINICAL TRIAL: NCT02660970
Title: Comparison of the Therapeutic Effect of Acupressure Therapy and Iberogast ® (STW-5) in Children With Functional Nausea - a Randomized Clinical Trial With Sham-conditions
Brief Title: Comparison of the Therapeutic Effect of Acupressure Therapy and Iberogast ® (STW-5) in Children With Functional Nausea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EKNZ 2015-322
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Functional Nausea
Keywords: Iberogast; Acupressure; gut-brain-axis
MeSH Terms: interventions — Acupressure; iberogast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Acupressure (Active Comparator): Children will have to wear a 'seasickness-band', which has the effect of acupressure
  Interventions: Other: Acupressure
- Placebo-band (Placebo Comparator): Children will have to wear a 'placebo-wristband'
  Interventions: Other: Placebo-band
- Iberogast (Active Comparator): Children will have to take Iberogast drops
  Interventions: Drug: Iberogast
- Placebo-drops (Placebo Comparator): Children will have to take placebo-drops
  Interventions: Other: Placebo-drops

INTERVENTIONS:
Other: Acupressure — Children will have to wear a 'seasickness-band', which has the effect of acupressure
  Other Names: Seasickness-Band
  Arms: Acupressure
Other: Placebo-band — Children will have to wear a 'placebo-wristband'
  Arms: Placebo-band
Drug: Iberogast — Children will have to take Iberogast drops
  Arms: Iberogast
Other: Placebo-drops — Children will have to take placebo-drops
  Arms: Placebo-drops

SUMMARY:
Functional gastrointestinal disorders are common disorders that are characterized by persistent and recurring GI symptoms. These occur as a result of abnormal functioning of the GI tract and are not caused by structural or biochemical abnormalities. As a result, medical tests- such as blood tests and endoscopic exams- have essentially normal/negative (non-disease) results. More than 20 functional GI disorders have been identified. They can affect any part of the GI tract. One of the most common functional disorders is nausea and dyspepsia (pain or discomfort in the upper abdominal area, feeling of fullness, bloating). Any chronic illness, including functional nausea, will affect a person's health-related quality of life (general well-being, ability to carry out everyday activities), additional psychosocial disturbances and amplify the experienced illness.

The majority of children suffering from functional nausea in Europe are treated with Iberogast®. a herbal mixture, whose effect was demonstrated in several studies. Since Iberogast® is not available in the United States of America, children there receive an acupressure therapy. The American gastroenterologists refer hereby to several studies, which have shown, that the positive effect of such therapies in patients with chemotherapy-induced nausea is even greater than a therapy with ondansetron. Since acupressure is able to reduce somatic nausea, it is also believed to decrease functional nausea, but it has never been investigated. Therefore, there are no data. That's why Investigators want to compare the efficacy of these two therapies, that is, Iberogast® and acupressure

DETAILED DESCRIPTION:
Functional gastrointestinal disorders are common disorders that are characterized by persistent and recurring GI symptoms. These occur as a result of abnormal functioning of the GI tract and are not caused by structural or biochemical abnormalities. As a result, medical tests- such as blood tests and endoscopic exams- have essentially normal/negative (non-disease) results. More than 20 functional GI disorders have been identified. They can affect any part of the GI tract. One of the most common functional disorders is nausea and dyspepsia (pain or discomfort in the upper abdominal area, feeling of fullness, bloating). Any chronic illness, including functional nausea, will affect a person's health-related quality of life (general well-being, ability to carry out everyday activities), additional psychosocial disturbances and amplify the experienced illness.

However, the majority of children suffering from functional Nausea in Europe get treated with Iberogast®: A herbal mixture, whose effect was demonstrated in several studies [10, 11]. Since Iberogast® is not available in the United States of America, children receive there an acupressure therapy. The American gastroenterologists refer hereby to several studies, which have shown, that the effect of such therapies in patient with chemotherapy-induced nausea is even greater than the taking of ondansetron [12,13 ]. Since acupressure is capable to reduce somatic nausea, it is also believed to decrease functional nausea, but it has never been investigated, therefore no data are available. That's why Investigators plan to compare the efficiency of these two therapies.

Furthermore Investigators want to measure the cognitive performance before and after the intervention to proof a possible effect on the 'gut-brain-axis'. For this purpose the participants have to do the 'Flanker Task', a standardised test on the computer.

ELIGIBILITY:
Inclusion Criteria:

* Functional nausea (normal endoscopy findings)

Exclusion Criteria:

* Gastrointestinal infection less than 2 weeks ago
* Known chronic gastrointestinal disease
* Use of drugs 2 weeks prior to starting the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
comparison in the levels of nausea as assessed by visual analog scales (VAS) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Furlano, MD, Dr, Principal Investigator — University Children's Hospital
Locations (1):
- Department of Pedriatric Gastroenterology, University Children's Hospital Basel, Basel, Canton of Basel-City, Switzerland